CLINICAL TRIAL: NCT04441970
Title: The Influence of Head and Neck Position on the Cuff Pressure Using Nasotracheal Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4-2020-0442
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Adult Patients Over 20 Years of Age Who Require Intubation of the Nasotracheal Tube to Undergo Oral and Maxillofacial Surgery Under General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neutral position (Active Comparator): General anesthesia will be induced and nasotracheal tube will be placed through the patient's nose. After 30 seconds, the cuff pressure will be measured using a cuff manometer. Inspiratory tidal volume, expiratory tidal volume, peak inspiratory pressure, and end-tidal carbon dioxide waveform will be recorded three times according to breathing. Whether ventilation is not adequate and air is leaking will be recorded.
  Interventions: Procedure: Neutral position
- Head extension position (Experimental): After changing the posture of the head and neck into head extension, cuff pressure will be recorded.
  Interventions: Procedure: Head extension position
- Head flexion position (Experimental): After changing the posture of the head and neck into head flexion, cuff pressure will be recorded.
  Interventions: Procedure: Head flexion position
- Head rotation position (Experimental): After changing the posture of the head and neck into head rotation, cuff pressure will be recorded.
  Interventions: Procedure: Head rotation position

INTERVENTIONS:
Procedure: Neutral position — The cuff pressure will be recorded at the neutral head position.
  Arms: Neutral position
Procedure: Head extension position — The cuff pressure will be recorded at the head extension position.
  Arms: Head extension position
Procedure: Head flexion position — The cuff pressure will be recorded at the head flexion position.
  Arms: Head flexion position
Procedure: Head rotation position — The cuff pressure will be recorded at the head rotation position.
  Arms: Head rotation position

SUMMARY:
Nasotracheal tube is a commonly used for securing airways when performing general anesthesia in various oral and maxillofacial surgery such as tooth extraction, maxillary and mandibular fractures. After the nasotracheal tube is placed in the patient's trachea, the process of inflating the cuff at the end of the tube with air is required. If the cuff is inflated with excess air, the cuff may press the mucous membrane on the inner wall of the trachea, causing ischemia. Previous studies have shown that if the pressure in the cuff exceeds 30 cmH2O, it is highly likely to cause ischemia. In addition, it was found that the pressure in the excessively inflated cuff was associated with post-operative sore throat, vocal cord paralysis, and nerve damage. Moreover, the pressure in the cuff may vary according to the patient's head and neck posture. The pressure changes in the cuff may vary depending on the material and shape of the cuff. Therefore, we will investigate to evaluate the effect of head and neck posture on the pressure in the cuff of nasotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 20 years of age
* patients who require intubation of the nasotracheal tube to undergo oral and maxillofacial surgery under general anesthesia

Exclusion Criteria:

* Patients whose neck cannot be rotated due to cervical diseases, cervical fractures, and previous cervical surgery
* Patients undergoing emergency surgery
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
cuff pressure of the nasotracheal tube | for 10 minutes after intubating the nasotracheal tube. At Day 0.
  Cuff pressure will be measured in the various head and neck positions.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No